CLINICAL TRIAL: NCT02647619
Title: A Randomized Controlled Trial (RCT) Comparing Clostridium Histolyticum With Needle Aponeurotomy.
Brief Title: Dupuytren´s Disease Study. Primary Disease, MCP Joint, Xiapex, PNF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Ingi Thor Hauksson, MD, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2639063; 2013-001221-13 (EudraCT Number)
Record Dates: First submitted 2015-12-29; First posted 2016-01-06 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Dupuytren Contracture
Keywords: Primary Dd disase; MCP joint
MeSH Terms: conditions — Dupuytren Contracture | interventions — xiapex; Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Needle aponeurotomy (Active Comparator): percutaneous transection or pretendinous palmar dupytren cord
  Interventions: Procedure: Needle aponeurotomy
- Xiapex (Active Comparator): Injection of 0.58 mg collagenase into pretendinous palmar dupytren cord
  Interventions: Drug: Xiapex

INTERVENTIONS:
Drug: Xiapex — Injection of collagenase of primary dupytren cord
  Other Names: Xiaflex
  Arms: Xiapex
Procedure: Needle aponeurotomy — 26 G needle multiple perforation tecqnique with local anesthetic
  Other Names: Percutaneous needle fasiotomy
  Arms: Needle aponeurotomy

SUMMARY:
Aim:

Clinical RCT comparing functional results and recurrence rate following enzymatic treatment vs. needle aponeurotomy.

Materials and methods:

30° or more contracture of only one metacarpophalangeal (MCP) joint contracture of one of the three ulnar digits and less than 20° for the adjacent proximal interphalangeal (PIP) joint. Patients with primary disease of the hand. Total of 80 patients needed to detect difference of 13.5°.

1) Needle aponeurotomy 2) Clostridium Histolyticum treatment. Clinical follow ups 1,4 weeks, 16 weeks and 1,2 and 5 years. Functional outcome scores: URAM, Quick Dash, EQ5D, brief MHQ, VAS pain and VAS patient satisfaction. Total passive extension contracture reduction, recurrence rate and registration of complications.

DETAILED DESCRIPTION:
Open surgery (fascieectomy) has traditionally been considered the gold standard of treatment for Dupytren´s disease (Dd) despite considerable risk of complications.

There is an increasing interest in Scandinavia in the treatment of Dd with Clostridium Histolyticum (Xiapex ®, Auxillium). However the enzyme is expensive and long-term effects are not well documented. More studies are needed to analyze both short and long term clinical outcome as well as cost-benefit analysis.

The treatment arm of Xiapex in this study follows the recommendation as by the producer.

The other treatment of Dd contracture in this study is needle fasiotomy/aponeurotomy. We use multiple perforation technigue with 26 G needle needle, with as little local anesthesia (xylocin w adrenaline) as needed during contionus extension of the finger untill successfully extended.

The two procedures leave little scar tissue lessening the challenges posed by the reoperations.

Recurrence rate of contracture following different treatments of Dupuytren's disease differs widely in the literature, and the rate is influenced by multiple factors.

ELIGIBILITY:
Inclusion Criteria:

* Primary Dd disease (no earlier treatment for this condition of the hand involved)
* Single digit involvement, one of the three ulnar digits
* Average norwegian language skills.
* MCPJ contracture of 30 degrees or more and less than 20 degree involvement of the adjacent PIPJ
* Minimum 18 y.o.

Exclusion Criteria:

* Involvement of 2 fingers/joints
* Earlier treatment for Dd disease of the same hand, affection of addjecent PIPJ of 20 degrees or mor
* Pregnancy
* Ongoing treatment with platelet inhibitors
* Treatment with tetracycline 2 weeks prior to treatment date
* Poor norwegian language skills
* Participation in other studies 4 weeks prior or after treatment date
* "Need to treat" of both hands

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Reduction in Total Passive Extension Deficit | 5 years

SECONDARY OUTCOMES:
Quick Dash (Disabilities of the shoulder and Hand) | 5 years
EQ5D (Euroqol 5 Dimensions) | 5 years
Brief MHQ (Michigan Hand Questionare) | 5 years
URAM (Unité Rhumatologique des Affections de la Main) | 5 years
Jamar grip strength | 1,4,26 weeks and one year.
VAS (Visual analogue scale) pain | 1,4,26 weeks and one year
  0 is no pain, 10 maximum pain
VAS (Visual analogue sale) satisfaction | 1,4,26 weeks. 1,2 and 5 years
  0 is not satisfied, 10 maximum satisfied
Complications | 1,4,weeks One year
  AE,SAE,SUSAR
Recurrence | 1,4,26 weeks. 1,2 and 5 years
  def. 30 degrees of treated MCP joint, or 20 or more degrees of adjecent PIPJ

CONTACTS AND LOCATIONS:
Overall Officials: Per-Henrik Randsborg, PhD, Study Director — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Oslo, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No